CLINICAL TRIAL: NCT02704715
Title: Postoperative Pain of General Anesthesia in Orbital Disease and Ocular Tumor
Brief Title: Postoperative Pain in Orbital Disease and Ocular Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2016MEKY006
Record Dates: First submitted 2016-02-25; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; general anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- general anesthesia,orbital operation (Other): 1. diagnosed as orbital disease and ocular tumor
  2. over 16 years old
  3. orbital operation under general anesthesia
  Interventions: Procedure: general anesthesia,orbital operation

INTERVENTIONS:
Procedure: general anesthesia,orbital operation — to evaluate the pain under general anesthesia

SUMMARY:
The purpose of this study is to evaluate the postoperative pain after general anesthesia of orbital diseases and ocular tumor patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patients diagnosed of orbital diseases or ocular tumor over 16 years old of the postoperative pain after general anesthesia , and to analyze the related factors of pain after operation.

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old
* diagnosed as orbital disease or ocular tumor
* surgery under general anesthesia

Exclusion Criteria:

* any uncontrolled clinical problems

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
pain | 24 hours after surgery
  numerical rating scale, NRS will be used to measure the pain

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Master, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided